CLINICAL TRIAL: NCT07369752
Title: Enhancing Brain And Mental Health Through Breathing Practice: Clinical Applications In Rural Adolescents With Psychiatric Symptoms (Breathing Study ?Adolescent)
Brief Title: Enhancing Brain And Mental Health Through Breathing Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Pravesh Sharma, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-012922
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder; Anxiety; Adolescent
Keywords: Seokmun Hoheup; breathing
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rural adolescent patients (Experimental): Rural adolescent patients of Mayo Clinic Health Systems, aged 12 to 17 years, with a clinical diagnosis of mild to moderate anxiety and/or depression will follow a structured breathing practice (Seokmun Hoheup) at least 3 times per week.
  Interventions: Behavioral: Breathing Intervention

INTERVENTIONS:
Behavioral: Breathing Intervention — Participants will follow a structured breathing practice (Seokmun Hoheup) that progresses in incremental steps, beginning with 15 minutes, increasing to 30 minutes, and then to 36 minutes per session over the course of the program.

SUMMARY:
The purpose of this study is to evaluate the feasibility of a structured breathing intervention in rural adolescents diagnosed with anxiety and depression, recruited from outpatient pediatric and child/adolescent psychiatry clinics.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 12 and 17 who have been diagnosed with a major depressive disorder (mild or moderate) and/or an anxiety disorder.
* Participants may have co-occurring mild to moderate alcohol or drug use problems, provided these do not require immediate specialized treatment or crisis intervention.
* All participants must be receiving care at one of two participating MCHS outpatient psychiatry clinics and must reside in rural area (RUCA code 4-10).
* Participants must be able to read and understand English, and both parental or guardian consent and adolescent assent will be required.

Exclusion Criteria:

* Current suicidal ideation or self-harm behavior requiring immediate clinical intervention
* Presence of severe psychiatric comorbidities such as psychosis, bipolar disorder, depression with psychotic features, severe alcohol and drug use, or eating disorders.
* Participants with significant cognitive impairment that would interfere with study participation.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) score | 4 months
  The Feasibility of Intervention Measure (FIM) is a self-reported questionnaire for participants to rate the feasibility of the breathing practice intervention on a 5-point Likert scale. Possible scores range from 0 (Completely Disagree) to 5 (Completely Agree)
Acceptability of Intervention Measure (AIM) score | 4 months
  The Acceptability of Intervention Measure (AIM) is a self-reported, 4 question survey, for participants to rate their acceptance of the breathing practice intervention on a 5-point Likert scale. Possible scores range from 0 (Completely Disagree) to 5 (Completely Agree)
Intervention Appropriateness Measure (IAM) score | 4 months
  The Intervention Appropriateness Measure (IAM) is a self-reported, 4 question survey, for participants to rate the appropriateness of the breathing practice intervention on a 5-point Likert scale. Possible scores range from 0 (Completely Disagree) to 5 (Completely Agree)
Recruitment feasibility | 4 months
  Proportion of eligible adolescents enrolled out of total participants screened
Retention feasibility | 4 months
  Proportion of participants retained through final assessment out of total enrolled

SECONDARY OUTCOMES:
System Usability Scale (SUS) score | 4 months
  Digital usability will be assessed using the System Usability Scale (SUS) tool, a self-reported 10 question survey, for participants to rate the usability of the digital app platform on a 5-point Likert scale. Possible scores range from 0 (Completely Disagree) to 5 (Completely Agree)
Total number of log-ins | 4 months
  Total number of times participants logged into the digital app platform
Completion rate of assigned breathing practices | 4 months
  Adherence to breathing practice and intervention engagement will be assessed as the completion rate of assigned sessions as measured by the session attendance logs

OTHER OUTCOMES:
Feasibility of collecting physiological data from baseline to 4 months | Baseline to 4 months
  Feasibility will be assessed based on data completeness, participant tolerance, and procedural viability from those undergoing fNIRS or MRI testing.
Feasibility of collecting psychological data | Baseline to 4 months
  Feasibility will be assessed by focusing on data completeness of validated mental health measures to include GHQ, GAD, PHQ-9.

CONTACTS AND LOCATIONS:
Overall Officials: Pravesh Sharma, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Health System-Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials